CLINICAL TRIAL: NCT06801223
Title: A Multicenter, Open-label, Phase 1b Study to Assess the Pharmacokinetics, Safety, and Tolerability of Sulbactam-Durlobactam in Hospitalized Pediatric Patients From Birth to <18 Years Who Are Receiving Systemic Antibiotic Therapy for Suspected or Confirmed Acinetobacter Baumannii-calcoaceticus Complex Infection
Brief Title: A Study to Assess Sulbactam-durlobactam in Pediatric Patients With Acinetobacter Baumannii-calcoaceticus Complex Infection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innoviva Specialty Therapeutics (Industry)
Collaborators: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS2514-2023-002
Record Dates: First submitted 2025-01-16; First posted 2025-01-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acinetobacter Baumannii-calcoaceticus Complex Infection (ABC)
Keywords: Acinetobacter baumannii-calcoaceticus complex infection; Sulbactam-durlobactam; Hospital-acquired bacteria pneumonia; Ventilator-associated bacterial pneumonia; Acinetobacter; ABC infection
MeSH Terms: interventions — Sulbactam; durlobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Pediatric patients 12 years to <18 years of age
  Sulbactam 25mg/kg -Durlobactam 25mg/kg, not to exceed 1g sulbactam - 1g durlobactam (Every 6 hours)
  Interventions: Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 6 hours)
- Cohort 2 (Experimental): Pediatric patients 6 years to <12 years of age
  Sulbactam 25mg/kg -Durlobactam 25mg/kg, not to exceed 1g sulbactam - 1g durlobactam (Every 6 hours)
  Interventions: Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 6 hours)
- Cohort 3 (Experimental): Pediatric patients 1 year to <6 years of age
  Interventions: Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 6 hours)
- Cohort 4 (Experimental): Pediatric patients 3 months to <1 year of age
  Interventions: Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 6 hours)
- Cohort 5 Subgroup 1 (Experimental): Aged 2 months to <3 months, term and preterm (gestational age >28 weeks)
  Term infants will receive 25mg/kg SUL and 25mg/kg DUR
  Preterm infants will receive 20mg/kg SUL and 20mg/kg DUR
  Interventions: Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 6 hours); Drug: Sulbactam 20mg/kg-Durlobactam 20mg/kg (Every 8 hours)
- Cohort 5 Subgroup 2 (Experimental): Aged birth to <2 months, term and preterm (gestational age >28 weeks and post-natal age >7 days)
  Term infants will receive 25mg/kg SUL and 25mg/kg DUR
  Preterm infants will receive 20mg/kg SUL and 20mg/kg DUR
  Interventions: Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 8 hours); Drug: Sulbactam 20mg/kg-Durlobactam 20mg/kg (Every 12 hours)

INTERVENTIONS:
Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 6 hours) — 25mg/kg SUL and 25mg/kg DUR
  Other Names: SUL-DUR
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5 Subgroup 1
Drug: Sulbactam 20mg/kg-Durlobactam 20mg/kg (Every 8 hours) — 20mg/kg SUL and 20mg/kg DUR
  Other Names: SUL-DUR
  Arms: Cohort 5 Subgroup 1
Drug: Sulbactam 25mg/kg -Durlobactam 25mg/kg (Every 8 hours) — 25mg/kg SUL and 25mg/kg DUR
  Other Names: SUL-DUR
  Arms: Cohort 5 Subgroup 2
Drug: Sulbactam 20mg/kg-Durlobactam 20mg/kg (Every 12 hours) — 20mg/kg SUL and 20mg/kg DUR
  Other Names: SUL-DUR
  Arms: Cohort 5 Subgroup 2

SUMMARY:
The goal of this clinical trial is to investigate the use of Sulbactam-Durlobactam (SUL-DUR) in pediatric patients and is being conducted to collect pharmacokinetic (PK) and safety data to enable the identification of appropriate pediatric dosing regimens for patients with Acinetobacter baumannii-calcoaceticus complex (ABC) infections

ELIGIBILITY:
Inclusion Criteria:

1. Patient from birth (defined as post-natal age of 7 days) to <18 years of age at the time of written informed consent (and assent, if applicable) and is hospitalized.
2. Patient and/or parent(s) or legal guardian(s) have provided the written informed consent and/or assent.
3. Patient has confirmed or suspected diagnosis of ABC infection and requires IV antibiotics for treatment.
4. Patient has expected survival of 30 days after enrollment in the study.
5. If patient is an individual of childbearing potential or reproductive potential, then the patient must remain abstinent OR must utilize one of the highly effective methods of contraception (ie, condom, combined oral contraceptive, implant, or injectable) from at least 30 days prior to screening until at least 30 days after administration of the last dose of study drug.

Exclusion Criteria:

1. Patient is a preterm infant, born at <28 weeks gestational age.
2. Patient has history of significant hypersensitivity or allergic reaction to any β-lactam, any contraindication to the excipients used in the formulation, or any contraindication to the use of β-lactam antibiotics. Note: For β-lactams, a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment.
3. Patient is in refractory septic shock at the time of enrollment, defined as persistent hypotension despite adequate fluid resuscitation or vasopressive therapy.
4. Patient is pregnant, breastfeeding, or intends to become pregnant.
5. Patient is receiving peritoneal dialysis or cardiopulmonary bypass.
6. Patient has planned blood transfusion within 24 hours of study drug administration and for the duration of the trial.
7. Patient is a newborn with clinically significant anemia who, in the opinion of the investigator, will not be able to tolerate the necessary blood draws to complete the study activities.
8. Patient (or patient's mother, if the patient is being breastfed) is using or will need to use any medications known to inhibit organic anion transporter 1 (OAT1) (eg, probenecid).
9. Patient has clinically significant renal, hepatic, or hemodynamic instability.
10. For Cohorts 1 through 3 only: patient has weight outside of the 5th to 95th percentile based on age.
11. Patient has an age-appropriate estimated creatinine clearance that indicates renal impairment.
12. Patient has the following laboratory results at Screening:

    1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3×upper limit of normal (ULN) and,
    2. Total bilirubin >2×ULN for age with conjugated/direct bilirubin >20% of the total. Note: Patients with AST or ALT up to 5×ULN are eligible if these elevations are acute and are documented as being directly related to the infectious process being treated.
13. Patient has clinically significant abnormal laboratory test results not related to the underlying infection that might expose the patient to risk by participating in the trial, confound the results of the trial, or interfere with the patient's participation for the full duration of the trial.
14. Patient (or patient's mother, if the patient is being breastfed) has participated in a clinical study involving investigational medication or an investigational device within the last 30 days or 5 half-lives, whichever is longer, prior to first dose of the study drug.
15. Patient has any condition that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the data.
16. Patient is unable or unwilling, in the opinion of the investigator, to comply with the protocol.
17. Patient (or patient's mother, if the patient is being breastfed) has previously received durlobactam.
18. Patient (or patient's mother, if the patient is being breastfed) has received sulbactam and/or sulbactam-containing regimens (eg, Unasyn) within 72 hours of first dose of the study drug.
19. Patient (or patient's mother, if the patient is being breastfed) has received amphotericin B within 7 days of first dose of the study drug.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-05-05 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Assess the pharmacokinetic (PK) parameters for maximum concentration (Cmax) of sulbactam and durlobactam | Day 1 and Day 3
Assess the PK parameters for area under the plasma concentration-time curve from 0 to 24 hours (AUC 0-24) of sulbactam and durlobactam | Day 1 and Day 3

SECONDARY OUTCOMES:
Percentage of participants experiencing Treatment Emergent Adverse Events (TEAEs) | 28 days
  Defined as any adverse event occurring after exposure to the study drug or any AE that worsens in intensity or frequency
Percentage of TEAEs leading to study drug discontinuation | 28 days
Incidence of related TEAEs | 28 days
Incidence of serious TEAEs | 28 days
Change from baseline values of liver function measured by Comprehensive Metabolic Panel (CMP) | Baseline and Day 28
Change from baseline values of kidney function measured by CMP | Baseline and Day 28
Change from baseline values of hemoglobin | Baseline and Day 28
Change from baseline value of white blood cell count | Baseline and Day 28
Change from baseline value of platelets | Baseline and Day 28
Change from baseline value of diastolic blood pressure | Baseline and Day 28
Change from baseline value of systolic blood pressure | Baseline and Day 28
Change from baseline values of heart rate | Baseline and Day 28
Change from baseline value of respiration rate | Baseline through Day 28
Change from baseline value of temperature | Baseline and Day 28

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Medical Center, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - ECU Brody School of Medicine, Greenville, North Carolina
  - University of Texas Medical Branch at Galveston, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests may be submitted starting 6 months after primary article publication and the data will be made accessible for up to 24 months; extensions may be considered on a case-by-case basis. Access criteria: Subject to certain criteria, conditions, and exceptions and upon completion of the review
Access Criteria: Subject to certain criteria, conditions, and exceptions and upon completion of the review and approval of the Research Proposal and Statistical Analysis Plan, Qualified Researchers engaging in independent scientific research can be provided de-identified IPD following the execution of a Data Sharing Agreement